CLINICAL TRIAL: NCT02475070
Title: Study of the Effect of Vildagliptin Versus Dapagliflozin on Glucagon Response to Mixed Meal in Metformin-treated Subjects With Type 2 Diabetes
Brief Title: Vildagliptin Versus Dapagliflozin on Glucagon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 350A
Record Dates: First submitted 2015-06-15; First posted 2015-06-18 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin first (Active Comparator): Treatment with vildagliptin 50mg twice daily for two weeks followed by four weeks washout and then treatment with dapagliflozin 10mg once daily for two weeks
  Interventions: Drug: Vildagliptin; Drug: Dapagliflozin
- Dapagliflozin first (Active Comparator): Treatment with dapagliflozin 10 mg once daily for two weeks followed by four weeks washout and then treatment with vildagliptin 50 mg twice daily for two weeks
  Interventions: Drug: Vildagliptin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin added at 50 mg twice daily for two weeks followed by four weeks washout and then dapagliflozin 10mg once daily for two weeks
  Other Names: Galvus
Drug: Dapagliflozin — Dapagliflozin added at 10 mg once daily for two weeks followed by four weeks washout and then vildagliptin 50 mg twice daily for two weeks
  Other Names: Forxiga

SUMMARY:
The aim of the study is to assess if vildagliptin and dapagliflozin have dissociated effects on glucagon secretion after a mixed meal ingestion in metformin-treated subjects with type 2 diabetes and whether this is associated with effects on glucose homeostasis.

DETAILED DESCRIPTION:
The aim of the study is to assess if vildagliptin and dapagliflozin have dissociated effects on glucagon secretion after a mixed meal ingestion in metformin-treated subjects with type 2 diabetes and whether this is associated with effects on glucose homeostasis. Subjects will therefore be treated with vildagliptin or dapagliflozin as add-on to metformin for two weeks followed by a meal test in which glucagon levels will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent has been given.
2. Patients with type 2 diabetes treated with a stable dose of metformin during the last three months
3. Age 20-70 years.
4. HbA1c 6.5-8.5% (48-67 mmol/mol) at visit 1.
5. Ability to complete the study

Exclusion Criteria:

1. Use of other glucose-lowering therapy than metformin within three months prior to visit 1.
2. A history of any secondary forms of diabetes, e.g., Cushing's syndrome and acromegaly.
3. Type 1 diabetes, positive GAD antibodies
4. Estimated glomerular filtration rate <60 ml/min
5. Acute infections which may affect blood glucose control within 4 weeks prior to visit 1
6. Any history of recent (<2 weeks) recurrent or severe hypoglycemic episodes.
7. Any history of acute pancreatitis
8. Any history of anaphylaxis, angioedema, and exfoliative skin conditions including Stevens-Johnson syndrome.
9. Liver disease such as cirrhosis or chronic active hepatitis
10. History of coronary heart disease or heart failure class III or IV
11. Donation of one unit (500 ml) or more of blood, significant blood loss equaling to at least one unit of blood within the past 2 weeks or a blood transfusion within the past 8 weeks.
12. Treatment with growth hormone of chronic oral or parenteral corticosteroid treatment (> 7 consecutive days of treatment) within 8 weeks prior to visit 1.
13. Use of other investigational drugs at visit 1 or within 30 days of visit 1, unsuitable for the study
14. Hypersensitivity to vildagliptin or dapagliflozin or any compound in the tablet core

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahren, MD PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Vildagliptin First: First intervention vildagliptin 50mg twice daily (2 weeks), Washout (4 weeks), Second intervention dapagliflozin 10mg once daily (2 weeks)
- Dapagliflozin First: First intervention dapagliflozin 10mg once Daily (2 weeks), washout (4 weeks), second intervention with vildaglipitn 50mg twice Daily (2 weeks)
Period: Overall Study
Arm/Group | Vildagliptin First | Dapagliflozin First
Started | 17 | 11
Completed | 17 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vildagliptin First | Dapagliflozin First | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (7.3) | 61 (6.7) | 63 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 11 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Glucagon Response to Meal
Description: Area under the curve (AUC) of the 180 min glucagon levels after mixed meal ingestion (0, 5, 10, 15, 30, 45, 60, 75, 90, 120, 150,180 and 240 minutes post-dose)
Time Frame: 240 min
Measure: Mean (Standard Error); unit: nmol/l min
Groups:
- Vildagliptin Treatment: Vildagliptin 50mg twice daily for 2 weeks
- Dapagliflozin Treatment: Dapagliflozin 10mg once Daily for 2 weeks
Arm/Group | Vildagliptin Treatment | Dapagliflozin Treatment
Number analyzed (Participants) | 28 | 28
nmol/l min | 39.0 (2.6) | 38.8 (2.7)

2. Secondary Outcome: Incretin Hormones
Description: Area under the curve (AUC) of the 180 min glucagon like peptide-1 levels after mixed meal (0, 5, 10, 15, 30, 45, 60, 75, 90, 120, 150, 180 and 240 minutes post-dose)
Time Frame: 240min
Measure: Mean (Standard Error); unit: nmol/l min
Arm/Group | Vildagliptin Treatment | Dapagliflozin Treatment
Number analyzed (Participants) | 28 | 28
nmol/l min | 3.8 (0.5) | 3.7 (0.5)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Vildagliptin: Treatment with vildagliptin 50mg twice daily for two weeks
- Dapagliflozin: Treatment with dapagliflozin 10 mg once daily for two weeks
Arm/Group | Vildagliptin | Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 4/28 | 5/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vildagliptin (N=28) | Dapagliflozin (N=28)
common cold (Infections and infestations) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Fatigue (Nervous system disorders) | 1 (1) | 1 (1)
Thirst (Metabolism and nutrition disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT02475070/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT02475070/SAP_001.pdf